CLINICAL TRIAL: NCT06965244
Title: Lenalidomide vs mEthotrexate in dIfficult-to-treat cutaneouS lUpus eRythEmatosus : An Assessor-blinded Randomized Clinical Trial
Brief Title: Lenalidomide vs Methotrexate in Difficult-to-treat Cutaneous Lupus Erythematosus
Acronym: LEISURE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP240920; 2024-520089-70-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-10; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Cutaneous Lupus Erythematosus (CLE)
Keywords: systemic lupus erythematosus; cutaneous lupus erythematosus; chronic CLE; lenalidomide; methotrexate; Resistance to anti-malarial
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Systemic | interventions — Lenalidomide; Methotrexate

STUDY DESIGN:
Intervention Model Description: The trial is a prospective, multicentre, randomised (1:1), open label, parallel group comparison with blinded assessment of the primary endpoint (PROBE design) conducted for comparing the efficacy and safety of lenalidomide 5 mg/day versus oral methotrexate 15 to 20 mg/week 16 for improving active CLE lesions for patients with isolated CLE or CLE.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lenalidomide with aspirin (Experimental): Lenalidomide with low-dose aspirin
  Interventions: Drug: Lenalidomide
- Methotrexate with folic acid (Active Comparator): Methotrexate with low dose of folic acid
  Interventions: Drug: Methotrexate (MTX)

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide with oral dose of 5 mg/day during 16 weeks associated with low-dose aspirin of 100 mg/day except for patients already receiving anticoagulant therapy
  Arms: Lenalidomide with aspirin
Drug: Methotrexate (MTX) — Methotrexate oral dose of 15 mg per week for individuals < 80 kg, and a dose of 20mg per week for those over 80 kg, along with an equal dose of folic acid supplementation given 48 hours after each dose
  Arms: Methotrexate with folic acid

SUMMARY:
Cutaneous lupus erythematosus (CLE) is a heterogeneous inflammatory autoimmune disease associated or not with systemic lupus erythematosus (SLE). Active CLE often cause pain/burning sensation and may lead to permanent visible scars and cicatricial alopecia, with psycho-social consequences/poor quality of life. First-line antimalarials (AMs) are recommended in CLE in addition to topical corticosteroids/tacrolimus with long-term response rate around 50%. Oral glucocorticosteroids (GCs) are recommended in addition to AMs for short term therapy in severe or widespread active CLE lesions. In non-responders to AMs and low-dose oral GCs, i.e., difficult-to-treat CLE, guidelines recommend the add-on of methotrexate as preferential second-line agent, with an overall efficacy of 50% in observational studies. Thalidomide has shown response rate of ≈90% in CLE in a meta-analysis of observational studies and is recommended as a second or third-line agent. However, potential severe adverse events (AEs) including teratogenicity, peripheral neuropathy and thromboembolic events limit its use.

Biological therapies including belimumab and anifrolumab, are approved only for patients with associated SLE (and not for those with isolated CLE). Their efficacy has been demonstrated as add-on therapy versus placebo but not versus a comparative drug. Moreover, efficacy of belimumab seems limited in difficult to-treat CLE and has not been assessed using validated tool, as the Cutaneous Lupus Erythematosus Disease Area and Severity (CLASI) Index. Anifrolumab seems interesting in CLE associated with SLE, but its use is limited by monthly intravenous infusions, high cost and unknown long-term AEs. Moreover, its efficacy in isolated CLE has not been assessed.

Lenalidomide is a thalidomide analogue with in vitro 1000 more potent immunomodulatory properties. It is recommended as a third-line treatment in France. With more than 60 treated patients, it showed excellent and rapid efficacy with an absence of drowsiness and peripheral neuropathy with a low-dose regimen of 5 mg/day. The use of lenalidomide was to date limited by its very high cost and its indications were restricted to haematological disorders. For note, the prevention of the higher risk of thromboembolism with lenalidomide requires the daily use of low-dose aspirin.

In France, a generic of lenalidomide is now available with a monthly cost of 2 euros, allowing a broad-scale assessment of its efficacy. Finally, lenalidomide might have a better efficacy than methotrexate.

We hypothesize that lenalidomide would be more efficacious than methotrexate in difficult-to-treat CLE patients with or without associated SLE. We assume that such trial would not be supported by pharmaceutical companies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of at least 18 years of age
2. Affiliated to the French social security
3. Able to provide written informed consent
4. Histologically-confirmed diagnosis of active CLE with or without associated SLE, either historical or at screening
5. CLASI-A score ≥ 8 at both screening and randomization
6. Active CLE despite

   * AMs agents used for at least 3 months and at stable dose for at least 30 days prior to randomization or previously documented discontinuation of AMs due to poor tolerability an/or side effect and/or
   * stable dose of GCs ≤15mg/day and/or
   * stable dose of topical corticosteroids (TCS) or topical tacrolimus for at least 30 days prior to randomization
7. Accepting monthly plasma pregnancy test and using adequate contraception for at least 4 weeks before and until 4 weeks following treatment

Exclusion Criteria:

1. Kidney function, liver function, cell blood count and infectious serology incompatible with receiving the study treatments, according to the SMPC of each drug.
2. Alcoholism (1/ no more than 10 standard drinks per week, 2/ no more than two standard drinks per day, and 3/ at least two alcohol-free days every week)
3. Ongoing cancer, including solid tumors and hematologic malignancies
4. Active severe SLE features including lupus nephritis, neuropsychiatric SLE, serositis, severe haematological features (autoimmune hemolytic anemia, idiopathic thrombocytopenic purpura) requiring high dose oral or IV GC and/or mycophenolate mofetil or cyclophosphamide
5. Medications:

   * Previous failure of methotrexate and lenalidomide prescribed for active CLE
   * Use of classical immunosuppressant drugs (mycophenolate mofetil, azathioprine), thalidomide, dapsone, retinoids, Janus Kinase inhibitors for CLE or SLE 4 weeks before screening
   * Use of biological therapy for CLE or SLE (including belimumab, rituximab, obinituzumab, ustekinumab, anifrolumab) 12 weeks before screening
6. Contraindication to use low-dose aspirin: salicylate hypersensitivity, salicylate-induced asthma, constitutional or acquired bleeding disorder, active gastroduodenal ulcer, or history of digestive bleeding.
7. Arterial or unprovoked venous thromboembolic events ≤ 5 years (for note antiphospholipid syndrome treated with vitamin K antagonist without thromboembolic events in the last 5 years or patients with positive antiphospholipid autoantibodies will NOT be excluded)
8. Pregnant women, breastfeeding or planning to become pregnant during the study treatment period and 1 month after the last dose of study treatment
9. Patients under legal protection and inability to comply with study requirement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who achieve decrease of at least 50% from baseline in the CLASI activity (CLASI-A) score | At week 16
  CLASI : Cutaneous LE disease Area and Severity Index

SECONDARY OUTCOMES:
Percentage of patients reaching CLASI-A 70 | At week 16
  CLASI : Cutaneous LE disease Area and Severity Index
Proportion of participants who achieve complete or almost complete response (CLASI-A 0-3) | At week 16
  CLASI : Cutaneous LE disease Area and Severity Index
Percentage of patients reaching CLASI-A 70 | At week 24
  CLASI : Cutaneous LE disease Area and Severity Index
Proportion of participants who achieve complete or almost complete response (CLASI-A 0-3) | At week 24
  CLASI : Cutaneous LE disease Area and Severity Index
Variation of Quality of life using DLQI | At week 16
  DLQI : Dermatology Life Quality Index
Variation of Quality of life using DLQI | At week 24
  DLQI : Dermatology Life Quality Index
SLE activity using SLEDAI | Up to 24 weeks
  SLEDAI : Systemic Lupus Erythematosus Disease Activity Index
SLE flare using SENELA-SLEDAI Flare Index (SFI) | Up to 24 weeks
  SELENA : Safety of Estrogens in Lupus Erythematosus National Assessment SLEDAI : Systemic Lupus Erythematosus Disease Activity Index
Variation of GCs dose | Between inclusion and week 24.
Variation of damage in each group using CLASI-D | At week 24
  CLASI : Cutaneous LE disease Area and Severity Index
Variation of damage in each group using CLASI-D | At week 16
  CLASI : Cutaneous LE disease Area and Severity Index
Rate of adverse events | Up to 24 weeks

IPD SHARING:
Plan to Share IPD: No